CLINICAL TRIAL: NCT03153514
Title: Obinutuzumab Containing Conditioning Regimen for CLL Patients and Patients With Richter's Transformation Requiring an Allogeneic Stem Cell Transplantation
Brief Title: Obinutuzumab Containing Conditioning Regimen for Patients With Poor Risk CLL or Richter's Transformation Requiring Allogeneic Stem Cell Transplantation
Acronym: CLLTX1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Prematurely terminated due to poor accrual
Sponsor: German CLL Study Group (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLLTX1; 2015-000568-32 (EudraCT Number); ML29747 (Other: Roche Pharma AG)
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2019-10

CONDITIONS: Chronic Lymphocytic Leukemia; Richter's Transformation
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obinutuzumab (Experimental): Obinutuzumab i.v.
  Cycle 1: in the peri-transplant and transplantation phase
  Cycle 2: if active disease and/or MRD positivity on day +60, +90, +180 or +270
  Interventions: Biological: Obinutuzumab

INTERVENTIONS:
Biological: Obinutuzumab — Obinutuzumab i.v.
  [Day 0 = day of stem cell transplant]
  Cycle 1: 100 mg (d -8), 900 mg (d -7), 1000 mg (d -1, +7, +14)
  Cycle 2: 1000 mg (d +1, +8, +15, +22)
  Other Names: GA-101; Gazyva

SUMMARY:
The primary objective of the study is to evaluate the feasibility, efficacy and safety of an obinutuzumab containing conditioning regimen for poor risk CLL patients and patients with Richter's transformation requiring an allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
CLL is the most common haematological malignancy in the western world. Though in the majority it behaves like a chronic disease with minimal impact on life expectancy, in around 15-20% of the patients it takes a very aggressive course. Patients who experience a high grade transformation, i.e., Richter's transformation also have a poor prognosis. Despite the advent of new therapeutic agents like Bcl-2 and BTK inhibitors which are revolutionising the outlook for this particular patient cohort, allogeneic stem cell transplantation is the only currently available therapy with the potential to cure. The non relapse mortality associated with this treatment is a major deterrent for physicians and patients alike to opt this intervention. We propose a trial to study the use of a B-cell depleting agent, obinutuzumab to simultaneously reduce tumour bulk control and offer GvHD prophylaxis in the peri-transplant setting and thereby analyse its impact on non relapse morbidity and mortality as well as maximum minimum residual disease (MRD) eradication. All patients with poor risk CLL (current EBMT criteria) and Richter's transformation with the best possible response to available therapies will be considered for the trial. Due to the poor disease control associated with peri-transplant T-cell depletion, obinutuzumab will be used instead of T-cell depleting agents as GvHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Have documented CLL according to iwCLL criteria
2. a) CLL requiring transplant according to the consensus statement 2014

   * Non-response or early relapse within 24 months after purine analogue combination therapy or treatment of similar efficacy plus high risk CLL TP53 deletion/mutation (del 17p-) and/or del 11 plus response to kinase inhibitors or other small molecules or
   * Non-response or early relapse within 24 months after purine analogue combination therapy or treatment of similar efficacy and refractory to or non-tolerating kinase inhibitors or other small molecules or b) Transformation of CLL to aggressive NHL (Richter's transformation) The CLL patients should have at least one therapy with the newer targeted agents such as BCL-2 inhibitors or BCR targeting agents. Both poor risk CLL patients and patients with Richter's transformation should achieve the best possible response defined as disease sensitivity measured as CR, PR or SD prior to transplant with an available salvage therapy
3. Availability of a suitable fully matched (10/10) sibling or unrelated donor
4. Must have an Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1.
5. Hematology values within the following limits unless cytopenia is caused by the underlying disease, i.e., no evidence of additional bone marrow dysfunction (e.g. myelodysplastic syndrome 2, hypoplastic bone marrow):

   * Absolute neutrophil count ≥ 1.0 x 109/L
   * Platelets ≥ 50 x 109/L and more than 7 days since last transfusion
6. Adequate liver function as indicated by a total bilirubin AST, and ALT ≤1.5 the institutional ULN value, unless directly attributable to the patient's CLL
7. Negative serological testing for hepatitis B (HBsAg negative and anti-HBc negative, patients positive for anti-HBc may be included if PCR for HBV DNA is negative and HBV-DNA PCR is performed every month until 1 year after last dosage of obinutuzumab), negative testing for hepatitis-C RNA and negative HIV test within 6 weeks prior to registration
8. 18 years of age or older but not older then 70 years
9. Able and willing to provide written informed consent and to comply with the study protocol procedures
10. Patient agrees to inform other physicians about study participation

Exclusion Criteria:

1. Previous allogeneic stem cell transplant
2. Known central nervous system (CNS) involvement
3. Patients with a history of confirmed PML
4. Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (left ventricular ejection fraction < 50%).
5. Organ dysfunction DLCO < 50%, TLC < 70%, FEV1 < 70% and or receiving supplementary oxygen, Inadequate renal function: Creatinine clearance < 50ml/min
6. Patients with active non-controlled infectious disease under treatment (no decrease of CRP or PCT) including active viral infection and active fungal infections with radiological progression despite treatment with Ambisome or active Triazole for more than a month
7. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies. Known sensitivity or allergy to murine products
8. Hypersensitivity to obinutuzumab or to any of the excipients such as for example Mannitol
9. Hypersensitivity to Fludarabine or hypersensitivity to both Treosulphan and Busulphan or any of the excipients of the used products
10. Hypersensitivity to both Ciclosporin A and calcineurin inhibitors or hypersensitivity to Mycophenolat-Mofetil or any of the excipients of the used products
11. Uncontrolled haemolytic anemia
12. Participation in another experimental drug trial (including chemotherapy, antibody treatment, kinase inhibitors, BCL2-antagonists or immunmodulatory agents) with start of the conditioning regimen/first obinutuzumab application.
13. Pregnant women and nursing mothers (a negative pregnancy test is required for all women of childbearing potential within 14 days before start of treatment)
14. Fertile men or women of childbearing potential unless:

    * Surgically sterile or ≥ 2 years after the onset of menopause
    * Willing to use two methods of reliable contraception including one highly effective (Pearl Index < 1) such as oral hormonal contraceptives, intrauterine device, sexual abstinence and one additional effective (barrier) while on study and maintained for up to 3 years after allogeneic transplantation or 18 months after the last dose of obinutuzumab therapy, whichever is longer
15. Vaccination with a live vaccine a minimum of 28 days prior to randomization
16. Prisoners or patients who are institutionalized by regulatory or court order or persons who are in dependence to the sponsor or an investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
PD-free rate | 12 months post-transplant
  Rate of patients free from disease progression (key efficacy endpoint)

SECONDARY OUTCOMES:
Minimal residual disease (MRD) negativity rate | days +60, +90, +180, +270 and months 12, 18 and 24 post-transplant
  Minimal residual disease negativity rate at different time points
Overall response rate (ORR) | 6 months post-transplant
  The overall response rate (ORR) is defined as the proportion of patients having achieved a CR/CRi, clinical CR/CRi or PR (including PR with lymphocytosis) as best response (according to the IWCLL guidelines (2008)) until and including the response assessment six months after transplantation (=number of patients with best response CR/CRi, clinical CR/CRi or PR (with or without lymphocytosis) divided by the number of the ITT population)
Progression-free survival (PFS) | up to month 24 post-transplant
  Time from the date of enrolment to the date of first occurrence of progression (determined using standard IWCLL guidelines) or death from any cause, whichever occurs first.
Event-free survival (EFS) | up to month 24 post-transplant
  Time from the date of enrolment to the date of first occurrence of progression (determined using standard IWCLL guidelines), death from any cause or initiation of subsequent treatment, whichever occurs first.
Overall survival (OS) | up to month 24 post-transplant
  Time from the date of enrolment to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Michael von Bergwelt-Baildon, Prof. Dr. med. Dr. rer. nat., Principal Investigator — University Hospital of Cologne
Locations (7):
- Germany (7):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsklinikum München, München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results of the study — https://pubmed.ncbi.nlm.nih.gov/34881358/